CLINICAL TRIAL: NCT00872001
Title: The Effect Of Acadesine On Clinically Significant Adverse Cardiovascular and Cerebrovascular Events In High-Risk Subjects Undergoing Coronary Artery Bypass Graft (CABG) Surgery Using Cardiopulmonary Bypass (Protocol No. P05633): RED-CABG Trial (Reduction in Cardiovascular Events by AcaDesine in Subjects Undergoing CABG)
Brief Title: The Effect Of Acadesine On Reducing Cardiovascular and Cerebrovascular Adverse Events In Coronary Artery Bypass Graft (CABG) Surgery (Study P05633 AM1)(TERMINATED)
Acronym: RED-CABG
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P05633; MK-8395 (Other: Product Identification Number); RED-CABG (Other: Protocol Abbreviation)
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Results first posted 2012-12-20 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Coronary Artery Bypass; Myocardial Infarction; Ventricular Dysfunction, Left; Stroke; Cardiopulmonary Bypass
MeSH Terms: conditions — Myocardial Infarction; Ventricular Dysfunction, Left; Stroke | interventions — acadesine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acadesine (Active Comparator): Acadesine intravenous (IV) infusion, plus cardioplegia solution with acadesine, and priming solution with acadesine in the heart lung machine during cardiopulmonary bypass (CPB)
  Interventions: Drug: Acadesine
- Placebo (Placebo Comparator): Normal saline, IV infusion, plus cardioplegia solution with added normal saline, and priming solution with added normal saline in the heart lung machine during CPB
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Acadesine — Acadesine 42 mg/kg diluted in normal saline to a total of 500 mL, delivered as an IV infusion over approximately 7 hours commencing within approximately 30 minutes before induction of anesthesia at a rate of 0.1 mg/kg/min (translating into 1.2 mL/min for a 500 mL solution). In addition, a 5 µg/mL cardioplegia solution of acadesine will be administered, and acadesine will be added to the priming solution (5 µg/mL) in the heart lung machine during CPB.
  Other Names: SCH 900395
  Arms: Acadesine
Drug: Normal Saline — Normal saline, 500 mL delivered as an IV infusion over approximately 7 hours commencing within approximately 30 minutes before induction of anesthesia at a rate of 1.2 mL/min for a 500 mL solution. In addition, standard cardioplegia solution with added normal saline will be administered, and placebo (normal saline) will also be added to the heart lung machine priming solution.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether acadesine is effective in reducing the cardiovascular and cerebrovascular adverse events in high-risk participants undergoing CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* A high risk participant undergoing non emergency CABG surgery requiring CPB and cardioplegia.
* Age: >=50 years
* At least one of the following risk factors:

  * Female (but not pregnant or lactating), or
  * History of prior CABG, or
  * History of myocardial infarction (MI), or
  * History of ischemic stroke, or
  * Left ventricular ejection fraction <=30%, or
  * Diabetes mellitus requiring insulin and/or antidiabetic agents.
* Significant coronary artery stenosis

Exclusion Criteria:

* Planned valve replacement, carotid artery or aortic surgery, distal coronary endarterectomy,surgical ablation for cardiac arrhythmia, or ventricular aneurysmectomy, alone or with CABG surgery (repair for mild to moderate mitral valve disease with concomitant CABG is not excluded).
* Planned or staged major surgery within 30 days of CABG surgery
* CABG surgery using intermittent aortic cross clamping without cardioplegia.
* Minimally invasive surgery (ie, without use of CPB).
* MI within 5 days prior to surgery.
* Pre-operative or planned intra operative/postoperative use of intra-aortic balloon pump (IABP), ventricular assist device (VAD), extra-corporeal membrane oxygenator (ECMO), or other mechanical hemodynamic assist device.
* History or presence of gout or uric acid nephrolithiasis.
* Serum creatinine >2 mg/dL (180 µmol/L).
* Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 x Upper Limit of Normal (ULN).
* Adenosine, aminophylline, nicotinic acid, pentoxifylline, theophylline, and any cardioplegia solution containing adenosine, dipyridamole or lidoflazine within 24 hours before surgery:
* Dipyridamole within 2 days and allopurinol or febuxostat within 4 days before surgery
* Food and drinks containing caffeine, theobromines or methylxanthines (such as coffee, tea, colas, some 'energy' drinks or chocolate) within 12 hours before surgery.
* Pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3080 (Actual)
Dates: Start 2009-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

REFERENCES:
- [Derived] Weisel RD, Nussmeier N, Newman MF, Pearl RG, Wechsler AS, Ambrosio G, Pitt B, Clare RM, Pieper KS, Mongero L, Reece TL, Yau TM, Fremes S, Menasche P, Lira A, Harrington RA, Ferguson TB; RED-CABG Executive and Steering Committees. Predictors of contemporary coronary artery bypass grafting outcomes. J Thorac Cardiovasc Surg. 2014 Dec;148(6):2720-6.e1-2. doi: 10.1016/j.jtcvs.2014.08.018. Epub 2014 Aug 14. PMID 25218533
- [Derived] Newman MF, Ferguson TB, White JA, Ambrosio G, Koglin J, Nussmeier NA, Pearl RG, Pitt B, Wechsler AS, Weisel RD, Reece TL, Lira A, Harrington RA; RED-CABG Steering Committee and Investigators. Effect of adenosine-regulating agent acadesine on morbidity and mortality associated with coronary artery bypass grafting: the RED-CABG randomized controlled trial. JAMA. 2012 Jul 11;308(2):157-64. doi: 10.1001/jama.2012.7633. PMID 22782417

RESULTS

PARTICIPANT FLOW:
Groups:
- Acadesine: Acadesine IV infusion, plus cardioplegia solution with acadesine, and priming solution with acadesine in the heart lung machine during cardiopulmonary bypass (CPB)
- Placebo (Normal Saline): Placebo (normal saline) IV infusion, plus cardioplegia solution with added normal saline, and priming solution with added normal saline in the heart lung machine during CPB
Period: Overall Study
Arm/Group | Acadesine | Placebo (Normal Saline)
Started | 1536 | 1544
Completed | 1400 | 1413
Not Completed | 136 | 131
Not completed — Adverse Event | 34 | 23
Not completed — Protocol Defined Clinical Event | 5 | 7
Not completed — Lost to Follow-up | 13 | 12
Not completed — Withdrawal by Subject | 18 | 30
Not completed — Protocol Violation | 5 | 8
Not completed — Did Not Meet Protocol Eligibility | 38 | 36
Not completed — Administrative | 23 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acadesine | Placebo (Normal Saline) | Total
Number analyzed (Participants) | 1536 | 1544 | 3080
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (8.5) | 66.7 (8.7) | 66.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 519 | 523 | 1042
  Male | 1017 | 1021 | 2038

OUTCOME MEASURES:

1. Primary Outcome: Incidence of All-cause Death, Non-fatal Stroke, and Need for Mechanical Support for Severe Left Ventricular Dysfunction (SLVD) (Intent-to-Treat Population)
Description: Incidence of all-cause death, non-fatal stroke, or need for mechanical support for SLVD (any component and composite) through post-operative Day 28 during and following CABG and administration of acadesine or placebo. Components defined as follows: All-cause death: Death from any cause, Non-fatal Stoke: occurrence of a stoke that was confirmed and adjudicated by Clinical Endpoints Committee that did not result in death, and Mechanical Support for SLVD: New use of any mechanical support for ≥1 hour for treatment of low cardiac output.
Time Frame: Up to Post-Operative Day 28
Population: The Intent-to-Treat Population included all participants randomly assigned to a treatment group and did not have to receive study drug. Each participant contributed to no more than one efficacy endpoint in any composite, i.e., a participant who experienced multiple components of an endpoint composite was counted only once in that composite.
Measure: Number; unit: Percentage of Participants
Groups:
- Placebo: Placebo (normal saline) IV infusion, plus cardioplegia solution with added normal saline, and priming solution with added normal saline in the heart lung machine during CPB.
Arm/Group | Acadesine | Placebo
Number analyzed (Participants) | 1536 | 1544
Percentage of Participants
  Composite of All Events | 4.9 | 4.9
  All-Cause Death | 1.9 | 1.7
  Non-Fatal Stroke | 1.7 | 1.7
  Need for Mechanical Support for SLVD | 2.2 | 2.3

2. Secondary Outcome: Incidence of Cardiovascular Death, Non-fatal Stroke, and Need for Mechanical Support for SLVD (Intent-to-Treat Population)
Description: Incidence of cardiovascular death, non-fatal stroke, and need for mechanical support for SLVD (any component and composite) through post-operative Day 28 during and following CABG and administration of acadesine or placebo. Components defined as follows: Cardiovascular death: Death due to cardiovascular causes, Non-fatal Stroke: occurrence of a stroke that was confirmed and adjudicated by Clinical Endpoints Committee that did not result in death, and Mechanical Support for SLVD: New use of any mechanical support for ≥1 hour for treatment of low cardiac output.
Time Frame: Up to Post-Operative Day 28
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Acadesine | Placebo (Normal Saline)
Number analyzed (Participants) | 1536 | 1544
Percentage of Participants
  Composite of All Events | 4.8 | 4.7
  Cardiovascular Death | 1.7 | 1.6
  Non-Fatal Stroke | 1.7 | 1.7
  Need for Mechanical Support for SLVD | 2.2 | 2.3

ADVERSE EVENTS:
Time Frame: Up to Post-Operative Day 28
Description: The As-Treated Population was used as the safety population and included all subjects who were assigned randomized treatment and received any amount of study drug (ie, acadesine or placebo).
Arm/Group | Acadesine | Placebo (Normal Saline)
Serious Adverse Events (participants affected / at risk) | 327/1442 | 329/1457
Other Adverse Events (participants affected / at risk) | 1154/1442 | 1189/1457
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acadesine (N=1442) | Placebo (Normal Saline) (N=1457)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Heparin-Induced Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 44 (46) | 41 (41)
Atrial Flutter (Cardiac disorders) | 2 (3) | 6 (6)
Atrial Rupture (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular Block Complete (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 4 (4) | 4 (4)
Cardiac Arrest (Cardiac disorders) | 12 (14) | 7 (8)
Cardiac Failure (Cardiac disorders) | 5 (5) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 11 (11) | 12 (13)
Cardiac Tamponade (Cardiac disorders) | 4 (4) | 4 (4)
Cardiac Valve Disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-Respiratory Arrest (Cardiac disorders) | 0 (0) | 4 (4)
Cardiogenic Shock (Cardiac disorders) | 4 (4) | 3 (4)
Cardiopulmonary Failure (Cardiac disorders) | 1 (1) | 1 (1)
Electromechanical Dissociation (Cardiac disorders) | 1 (1) | 2 (2)
Nodal Rhythm (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial Effusion (Cardiac disorders) | 2 (2) | 4 (4)
Right Ventricular Failure (Cardiac disorders) | 2 (2) | 0 (0)
Sick Sinus Syndrome (Cardiac disorders) | 4 (4) | 4 (4)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular Extrasystoles (Cardiac disorders) | 2 (2) | 2 (2)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricle Rupture (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular Extrasystoles (Cardiac disorders) | 3 (3) | 4 (4)
Ventricular Fibrillation (Cardiac disorders) | 5 (5) | 6 (6)
Ventricular Tachycardia (Cardiac disorders) | 3 (3) | 3 (3)
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 1 (1) | 0 (0)
Diabetic Retinopathy (Eye disorders) | 1 (1) | 0 (0)
Abdominal Adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis Ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestional Necrosis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 4 (4) | 5 (5)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 5 (5) | 4 (4)
Ileus Paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Ischaemia (Gastrointestinal disorders) | 4 (4) | 3 (3)
Intestinal Obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Large Intestine Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Malaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Oesophageal Spasm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Adverse Drug Reaction (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 4 (4) | 0 (0)
Catheter Site Haemorrhage (General disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 6 (6) | 1 (1)
Device Occlusion (General disorders) | 1 (1) | 0 (0)
Extravasation (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Gait Disturbance (General disorders) | 0 (0) | 1 (1)
General Physical Health Deterioration (General disorders) | 1 (1) | 0 (0)
Impaired Healing (General disorders) | 3 (3) | 1 (1)
Multi-Organ Failure (General disorders) | 4 (4) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1)
Organ Failure (General disorders) | 0 (0) | 1 (1)
Sudden Cardiac Death (General disorders) | 1 (1) | 0 (0)
Systemic Inflammatory Response Syndrome (General disorders) | 1 (1) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hydrocholecystis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactoid Reaction (Immune system disorders) | 1 (1) | 0 (0)
Abscess Limb (Infections and infestations) | 1 (1) | 0 (0)
Bacterial Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitus (Infections and infestations) | 5 (5) | 8 (8)
Cholecystitis Infective (Infections and infestations) | 0 (0) | 1 (1)
Clostridial Infection (Infections and infestations) | 1 (1) | 2 (2)
Drug Related Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1)
Haematoma Infection (Infections and infestations) | 0 (0) | 1 (1)
Incision Site Infection (Infections and infestations) | 3 (3) | 3 (3)
Infection (Infections and infestations) | 9 (9) | 9 (10)
Mediastinal Abscess (Infections and infestations) | 1 (1) | 1 (1)
Mediastinitis (Infections and infestations) | 2 (2) | 2 (2)
Pharyngitis Streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 10 (10) | 14 (14)
Postoperative Wound Infection (Infections and infestations) | 2 (2) | 2 (2)
Pyelonepritis (Infections and infestations) | 0 (0) | 1 (1)
Pyothorax (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 7 (7) | 6 (6)
Septic Shock (Infections and infestations) | 4 (4) | 2 (2)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal Mediastinitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 4 (4)
Wound Infection (Infections and infestations) | 6 (6) | 6 (6)
Wound Infection Pseudomonas (Infections and infestations) | 0 (0) | 1 (1)
Wound Infection Staphylococcal (Infections and infestations) | 0 (0) | 2 (2)
Collapse of Lung (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug Toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Graft Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision Site Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Operative Haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 16 (16) | 17 (17)
Postoperative Ileus (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Postoperative Renal Failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative Respiratory Distress (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Postoperative Thoracic Procedure Complication (Injury, poisoning and procedural complications) | 8 (8) | 3 (3)
Postpericardiotomy Syndrome (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Renal Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shunt Thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic Lung Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Graft Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vasoplegia Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weaning Failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Cardiac Output Decreased (Investigations) | 3 (3) | 0 (0)
Electrocardiogram Change (Investigations) | 1 (1) | 0 (0)
International Normalised Ratio Increased (Investigations) | 1 (1) | 0 (0)
Pulse Absent (Investigations) | 1 (1) | 0 (0)
White Blood Cell Count Increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid Overload (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Metabolic Disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fracture Delayed Union (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anoxic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular Incident (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Depressed Level of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 3 (3) | 0 (0)
Hypoxic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Paresis (Nervous system disorders) | 1 (1) | 0 (0)
Presynope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Affective Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination, Visual (Psychiatric disorders) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Transient Psychosis (Psychiatric disorders) | 1 (1) | 1 (1)
Acute Prerenal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 20 (21) | 14 (14)
Renal Failure Acute (Renal and urinary disorders) | 9 (10) | 10 (10)
Renal Tubular Necrosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3)
Acute Repiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 28 (31) | 26 (27)
Pleural Fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (4)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 12 (12)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Haematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory Alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 33 (34) | 23 (25)
Tracheal Stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Linear IGA Disease (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic Bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Incisional Drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Mechanical Ventilation (Surgical and medical procedures) | 3 (3) | 0 (0)
Thoracic Cavity Drainage (Surgical and medical procedures) | 0 (0) | 3 (3)
Air Embolism (Vascular disorders) | 1 (1) | 0 (0)
Aortic Rupture (Vascular disorders) | 1 (1) | 0 (0)
Arterial Thrombosis Limb (Vascular disorders) | 0 (0) | 1 (1)
Arteriovenous Fistula (Vascular disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 9 (9) | 5 (5)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Exsanguination (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haemodynamic Instability (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 14 (16) | 18 (18)
Jugular Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Labile Blood Pressure (Vascular disorders) | 0 (0) | 1 (1)
Lymphatic Fistula (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 2 (2) | 0 (0)
Peripheral Embolism (Vascular disorders) | 1 (2) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 2 (2) | 2 (2)
Peripheral Vascular Disorder (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Shock Haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis Superficial (Vascular disorders) | 1 (1) | 1 (1)
Venous Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
White Clot Syndrome (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acadesine (N=1442) | Placebo (Normal Saline) (N=1457)
Anaemia (Blood and lymphatic system disorders) | 384 (388) | 383 (387)
Leukocytosis (Blood and lymphatic system disorders) | 114 (117) | 95 (95)
Thrombocytopenia (Blood and lymphatic system disorders) | 119 (123) | 129 (129)
Atrial Fibrillation (Cardiac disorders) | 290 (303) | 328 (346)
Sinus Tachycardia (Cardiac disorders) | 81 (82) | 67 (67)
Constipation (Gastrointestinal disorders) | 207 (209) | 244 (245)
Nausea (Gastrointestinal disorders) | 354 (362) | 365 (373)
Vomiting (Gastrointestinal disorders) | 80 (81) | 86 (86)
Generalized Oedema (General disorders) | 87 (87) | 85 (85)
Oedema Peripheral (General disorders) | 108 (112) | 124 (134)
Pain (General disorders) | 100 (100) | 119 (123)
Pyrexia (General disorders) | 117 (122) | 105 (105)
Incision Site Pain (Injury, poisoning and procedural complications) | 218 (221) | 205 (211)
Procedural Pain (Injury, poisoning and procedural complications) | 560 (572) | 525 (543)
Hyperglycaemia (Metabolism and nutrition disorders) | 180 (181) | 165 (165)
Hypocalcaemia (Metabolism and nutrition disorders) | 85 (86) | 74 (74)
Hypokalaemia (Metabolism and nutrition disorders) | 139 (143) | 126 (127)
Anxiety (Psychiatric disorders) | 75 (75) | 88 (89)
Insomnia (Psychiatric disorders) | 89 (89) | 87 (87)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 257 (265) | 241 (252)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 323 (340) | 336 (352)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 59 (59) | 76 (76)
Hypertension (Vascular disorders) | 74 (76) | 74 (76)
Hypotension (Vascular disorders) | 280 (286) | 280 (283)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results

of the study without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication (including, without limitation, slides and texts of oral or other public presentations and texts of any transmission through any electronic media that report any study results).